CLINICAL TRIAL: NCT06893185
Title: Effectiveness of Cupping Therapy in Managing Neck Pain and Improving Cervical Mobility in Cervical Spondylosis Patients: A Randomized Clinical Trial
Brief Title: Cupping Therapy for Neck Pain in Cervical Spondylosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Dang Ngoc Ha Phuong, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 247/2024/HD-DHYD
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-04

CONDITIONS: Neck Pain; Cervical Spondylosis
Keywords: Neck Pain; Cupping therapy; Cervical spondylosis
MeSH Terms: conditions — Neck Pain; Spondylosis | interventions — Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dry cupping Group (Experimental): Dry cupping therapy every 3 days for a total of two weeks (5 sessions)
  Interventions: Other: Dry cupping therapy
- Electroacupuncture Group (Active Comparator): Electroacupuncture five times a week for a total of two weeks (10 sessions)
  Interventions: Other: Electroacupuncture

INTERVENTIONS:
Other: Dry cupping therapy — Dry cupping therapy will perform on the skin areas containing the EX-B2, A-shi, and GB21 acupuncture points every 3 days for 2 weeks.
  Arms: Dry cupping Group
Other: Electroacupuncture — Electroacupuncture therapy will be performed five times a week for 2 weeks. The acupoints are the Huatuojiaji (EX-B2), A-shi, and Jianjing (GB21).
  Arms: Electroacupuncture Group

SUMMARY:
Cervical spondylosis is one of the common causes of chronic neck pain. It can significantly affect the quality of life, lead to disabilities, and increase the economic burden on patients. Treatment mainly includes pain relievers, non-steroidal anti-inflammatory drugs (NSAIDs), muscle relaxants or physical therapy. The condition tends to recur frequently; therefore, long-term use of medication can lead to unwanted effects on the digestive system, kidneys, and cardiovascular system.

Dry cupping therapy is a non-pharmacological method that has been shown to be effective in pain management. Cupping therapy has the advantage of being applicable to patients who are afraid of needles and has a wide area of effect.

Given the limitations in evaluating treatment effectiveness and safety, along with the lack of published research discussing the analgesic effects of dry cupping for neck pain caused by cervical spondylosis, the investigators conducted the study on pain reduction and safety of cupping therapy in patients with neck pain caused by cervical spondylosis.

DETAILED DESCRIPTION:
Patients diagnosed with cervical spondylosis who have neck pain will be registered for this study. They will be treated with electroacupuncture or cupping therapy.

The intervention period is two weeks. Electroacupuncture will be performed five times a week while cupping therapy will be performed once every 3 days.

Data on the Visual Analog Scale (VAS) and side effects of electroacupuncture and cupping therapy will be recorded before the study and weekly for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 20 and 60 years, outpatient treatment.
* Individuals diagnosed with cervical spondylosis.
* Individuals report pain intensity between 3 and 8 according to on the Visual Analogue Scale (VAS) on the screening visit day.
* Experiencing neck pain for no longer than four weeks.
* Individuals who volunteered to participate in the study and signed a consent form.

Exclusion Criteria:

* Patients diagnosed with acute or chronic neck pain due to specific causes or with root compression syndrome, spinal cord compression syndrome, or vertebral artery syndrome.
* Patients loss of normal cervical curvature or deformity.
* Individuals with a history of neck trauma, cervical vertebra fracture, or cervical spine surgery, congenital spinal abnormalities, systemic bone and joint diseases.
* Patients have undergone cupping therapy, plastering, or drug inhalation within one week prior to participating in the study.
* Patients used of medications that could affect research outcomes within one week: Pain relievers, muscle relaxants, traditional medicines for treating neck pain.
* Patients suffer from a mental illness or lacks consciousness.
* Patients have a pacemaker, or any metal devices such as screws or plates.
* Patients currently using anticoagulant medications or has a bleeding disorder.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The change of the Visual Analog Scale (VAS) | Assessments were conducted before intervention and after each intervention week throughout the two weeks (Week 0, Week 1, Week 2)
  Symptom scores will be assessed based on a visual analogue scale (VAS). It usually consists of a 10 cm line anchored at each end by descriptors. Patients will be classified into 1 of 4 groups (no pain (0 cm), mild pain (1-3 cm), moderate pain (4-7 cm), severe pain (8-10 cm)).

SECONDARY OUTCOMES:
Proportion of intervention-related adverse events | Assessments were conducted after each intervention week throughout the two weeks.
  While dry cupping therapy and electroacupuncture is generally considered safe, some patients may experience minor side effects at the application site. These can include ecchymosis or burns. Rarely, more serious complications like dizziness, headaches, and fatigue may occur. The study will closely monitor and document any unexpected adverse events associated with the procedure.
Active range of motion of the cervical spine | Assessments were conducted before intervention and after each intervention week throughout the two weeks (Week 0, Week 1, Week 2)
  Active range of motion is measured using a goniometer. During measurement, the patient sits upright with hips and knees flexed at 90 degrees, both feet flat on the floor, and arms relaxed alongside the body. Cervical spine movements include flexion, extension, left and right lateral flexion, and left and right rotation.

REFERENCES:
- [Background] Kim S, Kim E, Jung G, Lee S, Kim JG. The hemodynamic changes during cupping therapy monitored by using an optical sensor embedded cup. J Biophotonics. 2019 May;12(5):e201800286. doi: 10.1002/jbio.201800286. Epub 2019 Jan 28. PMID 30604505
- [Background] Gao C, Wang M, He L, He Y, Li T. Alternations of hemodynamic parameters during Chinese cupping therapy assessed by an embedded near-infrared spectroscopy monitor. Biomed Opt Express. 2018 Dec 12;10(1):196-203. doi: 10.1364/BOE.10.000196. eCollection 2019 Jan 1. PMID 30775093
- [Background] Kolenkiewicz M, Wlodarczyk A, Wojtkiewicz J. Diagnosis and Incidence of Spondylosis and Cervical Disc Disorders in the University Clinical Hospital in Olsztyn, in Years 2011-2015. Biomed Res Int. 2018 Mar 25;2018:5643839. doi: 10.1155/2018/5643839. eCollection 2018. PMID 29770333
- [Background] Peng AT, Behar S, Yue SJ. Long-term therapeutic effects of electro-acupuncture for chronic neck and shoulder pain--a double blind study. Acupunct Electrother Res. 1987;12(1):37-44. doi: 10.3727/036012987816358922. PMID 2883835
- [Background] Zhang SP, Chiu TT, Chiu SN. Long-term efficacy of electroacupuncture for chronic neck pain: a randomised controlled trial. Hong Kong Med J. 2013 Dec;19 Suppl 9:36-9. PMID 24473589
- [Background] Chi LM, Lin LM, Chen CL, Wang SF, Lai HL, Peng TC. The Effectiveness of Cupping Therapy on Relieving Chronic Neck and Shoulder Pain: A Randomized Controlled Trial. Evid Based Complement Alternat Med. 2016;2016:7358918. doi: 10.1155/2016/7358918. Epub 2016 Mar 17. PMID 27073404
- [Background] Kim S, Lee SH, Kim MR, Kim EJ, Hwang DS, Lee J, Shin JS, Ha IH, Lee YJ. Is cupping therapy effective in patients with neck pain? A systematic review and meta-analysis. BMJ Open. 2018 Nov 5;8(11):e021070. doi: 10.1136/bmjopen-2017-021070. PMID 30397006
- [Background] Haldeman S, Carroll L, Cassidy JD. Findings from the bone and joint decade 2000 to 2010 task force on neck pain and its associated disorders. J Occup Environ Med. 2010 Apr;52(4):424-7. doi: 10.1097/JOM.0b013e3181d44f3b. PMID 20357682